CLINICAL TRIAL: NCT04179552
Title: Prospective, Open-label Clinical Investigation of Intra-articular Polyacrylamide Hydrogel Injection in Subjects With Knee Osteoarthritis
Brief Title: PAAG-OA Treatment for Knee Osteoarthritis
Acronym: IDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contura (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CON-OA
Record Dates: First submitted 2019-11-22; First posted 2019-11-27 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PAAG-OA (Experimental): All subjects receive treatment with PAAG-OA
  Interventions: Device: PAAG-OA

INTERVENTIONS:
Device: PAAG-OA — Intra-articular injection with PAAG-OA (polyacrylamide hydrogel)

SUMMARY:
This is a multi-centre, prospective, open-label, uncontrolled, clinical investigation followed by an open-label extension clinical investigation to evaluate PAAG-OA in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
This is a multi-centre, prospective, open-label clinical trial consisting of a main study followed by an extension study. The study will evaluate the effectiveness and safety of intra-articular polyacrylamide hydrogel (PAAG-OA) in subjects with knee OA.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged ≥ 18 years
4. Clinical diagnosis of knee OA according to American College of Rheumatology criteria
5. Definite radiographic OA in target knee at mild to severe stage (Kellgren-Lawrence 2-4)
6. Stable dose of analgesics for the past four weeks
7. Score of 2 or more (0-4 scale) on WOMAC question A1 (pain while walking on flat surface)
8. Body Mass Index (BMI) <35
9. For females of reproductive potential: use of adequate contraception must be used throughout the trial

Exclusion Criteria:

1. Female participants who are pregnant, lactating or planning pregnancy during the course of the clinical investigation
2. Previous intra-articular injection of polyacrylamide gel in the target knee
3. Previous intra-articular injection with hyaluronic acid or derivatives in target knee in the previous 6 months
4. Significant valgus/varus deformity of the knee, ligamentous laxity or meniscal instability
5. Diseases in target knee other than OA
6. Intra-articular injection of any substance other than hyaluronic acid (e.g. corticosteroids) in the target knee within the last 3 months
7. Acute serious infection of any region that required hospital care or intravenous antibiotic treatment within the last 30 days, or oral antibiotic treatment within the last 14 days
8. Skin disease or infections in the area of the injection site
9. History of sepsis in any joint or any clinical concern for an infectious process in the target knee
10. History of surgery in the target knee within the past 6 months
11. Symptomatic osteoarthritis of the hips, spine or ankle, that interferes with the evaluation of the target knee
12. Planned surgery on any lower extremity
13. Clinically significant venous of lymphatic stasis present in the legs
14. Suffering from any unstable or severe cardio-vascular disease
15. Any other contraindication to intra-articular injection
16. Any foreign material in the target joint
17. Any significant medical condition (e.g. significant psychiatric or neurological disorders or active alcohol/drug abuse) that is unstable/poorly controlled or other factors that may interfere with study participation
18. Treatment with systemic steroids with daily doses equivalent of >7,5 mg prednisolone
19. Significant change in physiotherapy in lower extremities related to OA within the previous month
20. Fibromyalgia
21. Inflammatory or other disease/condition which may affect the knee joint (e.g. rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis among others)
22. Haemophilia
23. Any other condition that in the opinion of the investigator puts a potential participant at risk or otherwise precludes participation in the investigation
24. Known allergic reactions to antibiotics (azithromycin and moxifloxacin) or local anaesthesia
25. Participation in any experimental device study within 6 months prior to enrolment, or participation in an experimental drug study within 1 month prior to enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Change in the WOMAC pain subscale | 3 months
  To evaluate the effectiveness of one injection of PAAG-OA on pain over 3 months in subjects with mild to severe knee OA. Change in WOMAC (WOMAC Osteoarthritis Index) pain subscale where a score of 0=none, and 4=extreme
WOMAC | 1 and 3 months
  To evaluate the effectiveness of one injection of PAAG-OA on knee OA-related subject reported symptoms, function during activities of daily living. Change in WOMAC (WOMAC Osteoarthritis Index) pain subscale where a score of 0=none, and 4=extreme
PGA | 1 and 3 months
  To evaluate the effectiveness of one injection of PAAG-OA on knee OA Patient Global Assessment (PGA). PGA is reported on a 10 cm Visual Analogue Scale

SECONDARY OUTCOMES:
Change in WOMAC | 6 and 12 months
  To evaluate the extended effectiveness of 6 ml PAAG-OA on knee OA-related subject reported symptoms, function during activities of daily living over 6 and 12 months. Change in WOMAC (WOMAC Osteoarthritis Index) pain subscale where a score of 0=none, and 4=extreme
Change in PGA | 6 and 12 months
  To evaluate the extended effectiveness of 6 ml PAAG-OA on knee OA-related Patient Global Assessment (PGA) over 6 and 12 months. PGA is reported on a 10 cm Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bliddal, MD, Principal Investigator — The Parker Institute
Locations (3):
- Denmark (3):
  - The Parker Institute, Frederiksberg
  - A2 Reumatologi og Idrætsmedicin, Hillerød
  - Reumatolog i Odense, Odense

REFERENCES:
- [Derived] Bliddal H, Hartkopp A, Beier J, Conaghan PG, Henriksen M. A prospective, open-label, clinical investigation of a single intra-articular polyacrylamide hydrogel injection in participants with knee osteoarthritis: a 5-year extension study. J Orthop Surg Res. 2025 Dec 12. doi: 10.1186/s13018-025-06526-0. Online ahead of print. PMID 41387884
- [Derived] Bliddal H, Beier J, Hartkopp A, Conaghan PG, Henriksen M. Effectiveness and safety of polyacrylamide hydrogel injection for knee osteoarthritis: results from a 12-month follow up of an open-label study. J Orthop Surg Res. 2024 May 2;19(1):274. doi: 10.1186/s13018-024-04756-2. PMID 38698396